CLINICAL TRIAL: NCT01358955
Title: A Multicenter, Randomized Trial to Assess Efficacy of Home-based and Group Cognitive Intervention Programs in Amnestic Mild Cognitive Impairment
Brief Title: Efficacy Study of Cognitive Intervention in Amnestic Mild Cognitive Impairment
Acronym: CogMCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inha University Hospital (Other)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Principal Investigator, Chul Soo Kim, Professor, Inha University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CogMCI study
Record Dates: First submitted 2011-05-20; First posted 2011-05-24 (Estimated); Last update posted 2013-08-28 (Estimated); Status verified 2013-08

CONDITIONS: Mild Cognitive Impairment
Keywords: mild cognitive impairment; cognitive therapy; prevention
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group cognitive intervention (Active Comparator): The cognitive training will be administered twice a week for 12 weeks, located in hospital-based outpatient memory clinics. Each session will last approximately 90 minutes. The cognitive training programs will be offered in group sessions consisted of 5 participants.
  Interventions: Other: group cognitive intervention
- Home-based cognitive intervention (Active Comparator): The participants will do their homework for 30 minutes every business days for 12 weeks.
  Interventions: Other: Home-based cognitive intervention
- Wait list Control (No Intervention): They will participate in cognitive intervention after ending this study.

INTERVENTIONS:
Other: group cognitive intervention — The cognitive training will be administered twice a week for 12 weeks, located in hospital-based outpatient memory clinics. Each session will last approximately 90 minutes. The cognitive training programs will be offered in group sessions consisted of 5 participants.
  Arms: Group cognitive intervention
Other: Home-based cognitive intervention — The participants will do their paper and pencil homework for 30 minutes every business days for 12 weeks.
  Arms: Home-based cognitive intervention

SUMMARY:
* There will be a significant difference in cognitive function between cognitive intervention group (group therapy) and a wait list control group.
* There will be a significant difference in cognitive function between a home-based cognitive intervention group and a wait list control group.

DETAILED DESCRIPTION:
The change of Modified ADAS-cog score from the baseline to post-intervention will be compared between the cognitive intervention group and wait list control group.

ELIGIBILITY:
Inclusion Criteria:

* 50 to 85 years of age
* memory complaint corroborated by a participant and an informant
* delayed recall score on the Seoul Verbal Learning Test (SVLT) below 1.0 standard deviations from the mean of the age and education-normative values among the Korean population
* Global CDR score is 0.5, Memory CDR score is 0.5 or 1.
* above 1.5 standard deviations from the mean of normative data of the respective age- and education-matched population on the Korean Mini-Mental State Examination
* normal functional activities
* not diagnosed with dementia
* Modified Hachinski Ischemic Score (HIS): 0-4
* brain magnetic resonance imaging or CT showing no clinical evidence of other diseases (i.e., normal pressure hydrocephalus, brain tumor, cerebrovascular disease) capable of producing cognitive impairment.
* Subjects are also required to have a reliable caregiver who meet the patient at least once a week and is sufficiently familiar with the patient to provide the investigator with accurate information.
* He/She can read and write
* written informed consent

Exclusion Criteria:

* any patient who were involved in other clinical trials or treated with experimental drug within 4 weeks
* any patients with any severe or unstable medical disease that may prevent the patient from completing all study requirements (i.e., unstable or severe asthma or cardiovascular disease, active gastric ulcer, severe hepatic or renal disease)
* any patients with clinically significant laboratory abnormalities such as an abnormal thyroid function test, abnormal low level of vitamin B12 or folate, or positive venereal disease research laboratory test
* any patients with any primary neurodegenerative disorder or psychiatric disorder other than AD (i.e., Parkinson's disease, schizophrenia, or major depressive disorder)
* any patients with any history of drug or alcohol addiction during the past 10 years
* any hearing or visual impairment that can disturb the efficient evaluation of the patient

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 293 (Actual)
Dates: Start 2011-03; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Modified Alzheimer's Disease Assessment Scale-Cognitive subscale(ADAS-cog) | postintervention, 12 weeks follow-up, and 24 weeks follow-up

SECONDARY OUTCOMES:
story recall test | postintervention, 12 weeks follow-up, and 24 weeks follow-up
Digit span forward and backward | postintervention, 12 weeks follow-up, and 24 weeks follow-up
Word fluency test | postintervention, 12 weeks follow-up, and 24 weeks follow-up
color-word stroop test | postintervention, 12 weeks follow-up, and 24 weeks follow-up
Digit symbol test | postintervention, 12 weeks follow-up, and 24 weeks follow-up
prospective memory test | postintervention, 12 weeks follow-up, and 24 weeks follow-up
Mini-Mental State Examination | postintervention, 12 weeks follow-up, and 24 weeks follow-up
CDR-SB | postintervention, 12 weeks follow-up, and 24 weeks follow-up
K-AD8 | postintervention, 12 weeks follow-up, and 24 weeks follow-up
PRMQ | postintervention, 12 weeks follow-up, and 24 weeks follow-up
MMQ-Strategy | postintervention, 12 weeks follow-up, and 24 weeks follow-up
QOL-AD | postintervention, 12 weeks follow-up, and 24 weeks follow-up
Geriatric Depression Scale-short form | postintervention, 12 weeks follow-up, and 24 weeks follow-up
Bayer ADL | postintervention, 12 weeks follow-up, and 24 weeks follow-up
CGA-NPI | postintervention, 12 weeks follow-up, and 24 weeks follow-up
Subjective cognitive assessment | postintervention, 12 weeks follow-up, and 24 weeks follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Seong H Choi, MD, PhD, Principal Investigator — Inha University Hospital
Locations (18):
- South Korea (18):
  - Korea University Medical College, Ansan
  - Soonchunhyang University Hospital, Bucheon-si
  - Bucheon St. Mary's Hospital, the Catholic University of Korea, Bucheon-si
  - Donga University Hospital, Busan
  - Pusan National University Hospital, Busan
  - Daejun Eulji University Hopistal, Daejun
  - Myongji Hospital, Goyang
  - NHIC Ilsan Hospital, Goyang
  - Inha Univeristy Hospital, Incheon
  - Jeju National University Hospital, Jeju City
  - Maryknoll Hospital, Pusan
  - Bobath Memorial Hospital, Seongnam
  - Sungkyunkwan University, Samsung Seoul Hospital, Seoul
  - Asan Medical Center, Psychiatry, Seoul
  - Inje University Sanggye Paik Hospital, Seoul
  - Konkuk University Medical Cener, Seoul
  - Ajou University Hospital, Suwon
  - Hyoja Geriatric Hospital, Yŏngin